CLINICAL TRIAL: NCT06778668
Title: Evaluation of the Effectiveness of Adding Fentanyl to Transversus Abdominis Plane Block in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effectiveness of Fentanyl-Added TAP Block in Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Mustafa Çabuk, Resident Doctor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UU-AN-MC-01
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into three groups:
  Group 1: TAP block with bupivacaine only, Group 2: TAP block with bupivacaine and fentanyl, Group 3: Control group (no TAP block).
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is a double-blind randomized trial. Both the researchers assessing postoperative pain and the participants will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Group 1, a unilateral TAP block will be applied using the linear probe (38 mm, 6 MHz) of the ultrasound device routinely used in our clinic. The procedure will be performed in the supine position under aseptic conditions. The ultrasound probe will be placed horizontally in the right subcostal region (an anatomical area following the lower border of the ribs). A 50 mm block needle will be advanced into the fascial plane between the transversus abdominis and rectus abdominis muscles. A total of 20 ml of 0.25% bupivacaine solution will be administered, with a maximum dose of 2 mg/kg.
  Interventions: Procedure: TAP block with bupivacaine only
- Group 2 (Active Comparator): In Group 2, a unilateral TAP block will be applied using the linear probe (38 mm, 6 MHz) of the ultrasound device in the supine position under aseptic conditions. The ultrasound probe will be placed horizontally in the right subcostal region, and a 50 mm block needle will be advanced into the fascial plane between the transversus abdominis and rectus abdominis muscles. A total of 20 ml of block solution containing 0.25% bupivacaine and 50 mcg fentanyl will be administered.
  Interventions: Procedure: TAP block with bupivacaine and fentanyl
- Group 3 (No Intervention): Patients in Group 3 will serve as the control group, and no block will be applied.

INTERVENTIONS:
Procedure: TAP block with bupivacaine only — Patients undergoing laparoscopic cholecystectomy will receive TAP block with bupivacaine only after induction and before the surgical procedure begins.
  Arms: Group 1
Procedure: TAP block with bupivacaine and fentanyl — Patients undergoing laparoscopic cholecystectomy will receive a TAP block with bupivacaine and fentanyl after induction and before the surgical procedure begins
  Arms: Group 2

SUMMARY:
The aim of this study is to evaluate the effectiveness of adding fentanyl to the TAP block in laparoscopic cholecystectomy cases. It is hypothesized that the addition of fentanyl to the TAP block will enhance the quality of postoperative analgesia and prolong the duration of blockade compared to the TAP block performed with bupivacaine alone. The study aims to determine the most effective approach by comparing these two treatment methods with a control group.

DETAILED DESCRIPTION:
Cholecystectomy was first performed in 1882 by Karl Langenbuch and is widely used for the treatment of symptomatic gallbladder diseases, such as acute cholecystitis and cholelithiasis. Today, the laparoscopic technique is preferred due to its advantages, including faster recovery, better cosmetic outcomes, and shorter hospital stays. However, despite these benefits, postoperative pain, particularly in the shoulder and abdomen, remains a common issue after laparoscopic surgery and is one of the primary causes of delayed discharge. This pain can be attributed to incision sites, peritoneal irritation caused by the insufflation gas, and trocar entry points.

Effective management of postoperative pain is crucial for accelerating recovery and preventing the development of chronic pain. One of the key strategies in multimodal analgesia is the Transversus Abdominis Plane (TAP) block, which can reduce both postoperative pain and the need for opioids. First described by Rafi in 2001, TAP block gained widespread use after Hebbart et al. demonstrated in 2007 that it could be applied more effectively and safely under ultrasound guidance. The block involves injecting local anesthetics into the neurofascial plane between the transversus abdominis and internal oblique muscles, where the intercostal, subcostal, ilioinguinal, and iliohypogastric nerves run.

Since the identification of opioid receptors in peripheral nerves, there has been interest in combining opioids with local anesthetics to enhance the duration and quality of peripheral nerve blocks. Studies have shown that certain opioids, including fentanyl and sufentanil, exhibit local anesthetic-like effects. Fentanyl, a commonly used opioid, has been shown to improve analgesia quality and prolong the duration of subarachnoid blocks when combined with local anesthetics.

This study aims to evaluate the effectiveness of adding fentanyl to the TAP block, which is routinely performed in our clinic, in laparoscopic cholecystectomy cases. The hypothesis is that the addition of fentanyl to bupivacaine in the TAP block will improve the quality of postoperative analgesia and prolong the block duration.

A total of 66 patients undergoing laparoscopic cholecystectomy will be included in the study. Patients will be randomized into three groups:

Group 1: TAP block with bupivacaine only, Group 2: TAP block with bupivacaine and fentanyl, Group 3: Control group (no TAP block). All patients will receive standard general anesthesia protocols, and TAP block will be performed before the surgical procedure. Postoperatively, pain scores (VAS), rescue analgesia requirements, additional analgesic and antiemetic use, complications, and patient satisfaction will be evaluated. The study will also assess whether fentanyl prolongs the block duration and improves postoperative analgesia quality.

The goal of this study is to compare these approaches and determine the most effective method for managing postoperative pain in laparoscopic cholecystectomy cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years
* American Society of Anesthesiologists (ASA) classification I-II-III according to the American Society of Anesthesiologists
* Patients who provide written informed consent
* Patients scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* Pregnancy or suspected pregnancy
* BMI > 35
* Known allergy to local anesthetics or opioids
* Suspected coagulopathy or infection at the injection site
* Severe neurological, psychiatric, cardiovascular, liver, or renal failure
* Patients converted to open surgery intraoperatively

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
The Visual Analog Scale | 1 day
  The Visual Analog Scale (VAS) is a simple and widely used tool to assess the intensity of pain or symptoms. It helps convert patients' subjective experiences (such as pain, discomfort, or fatigue) into a numerical value. This scale is particularly useful in evaluating postoperative pain and chronic pain conditions.
  How Does VAS Work? The VAS typically consists of a 10 cm horizontal or vertical line. One end of the line is labeled "No Pain", and the other end is labeled "Worst Pain Possible".
  The patient is asked to mark a point on the line that best represents their pain intensity.
  The marked point is measured with a ruler to obtain a score between 0 and 10.
  VAS Scoring:
  VAS Score Pain Level 0 No pain 1-3 Mild pain 4-6 Moderate pain 7-10 Severe and unbearable pain
  Areas of Use:
  Postoperative pain assessment Chronic pain management Conditions like migraine, arthritis, or cancer pain Evaluating physical and emotional symptoms (e.g., anxiety or depression)

SECONDARY OUTCOMES:
Rescue Analgesic Requirement | 1 day
  It will be applied to patients with a VAS score above 5.
The 5-point Likert scale | 1 day
  Patient satisfaction will be assessed using a 5-point Likert scale.The 5-point Likert scale is a widely used rating scale to measure attitudes, opinions, and perceptions in surveys and questionnaires. In clinical studies, it is often used to assess patient satisfaction, allowing patients to rate their experiences on a scale from strongly dissatisfied to strongly satisfied.
  Structure of the 5-Point Likert Scale:
  Score Response
  1. Strongly Dissatisfied
  2. Dissatisfied
  3. Neutral
  4. Satisfied
  5. Strongly Satisfied